CLINICAL TRIAL: NCT03173274
Title: Incentives to Promote Smoking Cessation in Low SES Women
Acronym: ProjectMIST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant funding ended for pilot work
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Rachel N Cassidy, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5-24001
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (CM) (Experimental): Those in the CM condition will continue to provide CO values twice-daily, and will receive escalating reinforcement values for CO values indicating continuous smoking abstinence (CO < 6 ppm).
  Interventions: Behavioral: Brief Motivational Intervention; Behavioral: Contingency Management
- Non-Contingent Reinforcement (Active Comparator): Participants in the NC condition will also provide CO levels twice-daily. However, their reinforcement will not be contingent upon their CO level but will be yoked to someone in the CM condition so that average reinforcer values are equivalent across the 2 conditions.
  Interventions: Behavioral: Brief Motivational Intervention; Behavioral: Non-Contingent Reinforcement

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — Participants in both groups will be given an BMI intervention in which they will be counseled to quit smoking.
Behavioral: Contingency Management — Contingent Reinforcement for negative breath CO samples
  Arms: Contingency Management (CM)
Behavioral: Non-Contingent Reinforcement — Participants will receive reinforcement for submitting samples ona yoked schedule unrelated to CO sample value [CM control]
  Arms: Non-Contingent Reinforcement

SUMMARY:
The purpose of this study is to investigate the feasibility of a mobile-phone based contingency management (CM) intervention for smoking in low-SES women. The CM intervention will be combined with a Brief Motivational Interviewing (BMI) counseling component. This study will examine the following research aims:

Primary Aim: To compare the effects of a Brief Motivational Intervention (BMI) + mobile phone-based CM on tobacco use when compared to BMI with a non-contingent control condition in a small feasibility trial.

Hypothesis: The investigators expect women in the BMI + CM condition to have more smoke free days than women in the BMI + NC condition.

Secondary Aim: To examine alcohol use as a moderator of cessation outcomes.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of preventable death in the United States, accounting for one out of every five deaths (CDC, 2012). In particular, smoking prevalence rates are high among socioeconomically-disadvantaged women; for example, over 40% of women with less than 12 yrs education smoke, compared to 28% and 16% among those with some college and undergraduate degrees (SAMHSA, 2010). Smoking cessation rates are particularly low among low-SES women with co-occurring alcohol use disorders, and these substances are frequently used together (Kahler et al., 2010; Businelle et al., 2013). Therefore, interventions that reduce both alcohol and smoking among heavy alcohol-using women are vitally needed to reduce rates of smoking-related morbidity and mortality in this vulnerable population.

Counseling approaches that incorporate problem solving, skills training and social support are effective for reducing smoking in the general population (Fiore et al., 2008). However, given the high rates of smoking among alcohol-using women, they may be inadequate for in this population. Contingency management (CM) interventions, which provide tangible reinforcers contingent upon smoking abstinence or reduction to a criterion level, are highly-efficacious interventions for reducing cigarette smoking and other drug use in low-SES women (Higgins et al., 2012). Within the theoretical framework of operant conditioning, increasing the availability of an alternative reinforcer weakens the amount of control that the drug has over the user's behavior, especially when obtaining the alternative reinforcer is contingent on behaviors incompatible with drug use (Higgins, 1997). The tenets of CM interventions include (1) arranging the environment such that the target behavior can be readily and objectively detected, (2) providing a tangible reinforcer when the target behavior occurs, and (3) withholding reinforcement when the target behavior does not occur (Higgins et al., 1994).

Although CM interventions clearly are effective at promoting smoking reductions, there are several challenges associated with translating CM into an effective clinical treatment for smoking. Perhaps the most significant challenge is the frequent monitoring necessary to objectively verify smoking abstinence using breath carbon monoxide (CO), the most convenient objective measure of smoking status. Because of the short half-life of CO (5-6 hours), CO levels must be measured at least twice per day in order to verify continuous abstinence. Recent CM-smoking studies have addressed this feasibility challenge by providing study participants with breath CO monitors and laptop computers or smartphones to use in their own natural environments (e.g., Dallery, Raiff & Grabinski, 2013). Participants are taught how to use their smartphones to text videos of themselves providing a breath CO level to a research staff member, twice per day. After the study staff has determined that the breath CO sample meets the abstinence criterion, participants are informed of the amount that they have earned for that sample.

Given the high rates of smoking in low-SES women, investigating the additive impact of an in-person brief counseling intervention and a phone-based CM intervention is an important next step in examining effective methods to reduce the impact of smoking in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Smoke an average of at least ten cigarettes per day for at least 1 year
* Breath CO levels > 8 ppm
* >12 years of education
* Reliable and consistent access to a smart phone with video messaging capabilities

Exclusion Criteria:

* Intention to quit smoking in the next 30 days
* Currently seeking treatment for smoking cessation.
* Currently using nicotine replacement therapies or other pharmacotherapies as cessation aid (intermittent use acceptable)
* No reliable access to a video-messaging smart phone
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
Percent of negative CO samples | End of two-week intervention
  The amount of negative, decreased CO samples submitted by participants

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No